CLINICAL TRIAL: NCT04685200
Title: Unraveling the Mechanisms Underlying Primary Sclerosing Cholangitis Through a Multidisciplinary, Integrative Research Approach
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000130; 000130-DK
Record Dates: First submitted 2020-12-24; First posted 2020-12-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-07-31

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Inflammatory Bowel Disease; Liver Disease; Natural History
MeSH Terms: conditions — Cholangitis, Sclerosing; Inflammatory Bowel Diseases; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: 90 controls to collect epidemiological data as well as blood samples, nasal swabs, salivary samples and stool samples from family members and cohabitants of subjects affected with PSC.
- PSC Pariticipants: 40 patients with PSC diagnosed by standard clinical, biochemical, or imaging features (including up to 30 with a known diagnosis of IBD)

SUMMARY:
Background:

Primary sclerosing cholangitis is a rare chronic liver disease. It affects the bile ducts of the

liver. It can result in bile duct infections, cirrhosis, cancer, and end stage liver disease. Researchers want to learn more about this disease.

Objective:

To understand the biological causes of primary sclerosing cholangitis.

Eligibility:

Adults age 18 and older who have primary sclerosing cholangitis.

Design:

Participants will be screened with a medical history, physical exam, and blood tests.

Participants will give blood, saliva, urine, and stool samples. They will have nasal swabs. They will complete surveys.

Participants will get an intravenous (IV) catheter. A plastic tube is inserted into an arm vein.

Participants will have a colonoscopy. A tube with a video camera at the end is inserted into the rectum.

Participants will have an upper endoscopy. A scope with a light and camera at its tip is used to look inside the upper digestive tract.

Participants will have a liver biopsy, entering through the chest wall or a neck vein. Blood is drawn from a blood vessel that carries blood to the liver. A liver tissue sample is taken.

Participants will have magnetic resonance imaging or spectroscopy. They will get a contrast agent through an IV.

Participants may have an optional bone marrow aspiration. A large needle is inserted into the hip to withdraw marrow.

Participants will have a liver ultrasound.

Participants will complete a 3-day food diary. They will have a nutrition assessment.

Participants may give contact details for people who live with them, to also take part in this study.

Participation will last for 12 months.

DETAILED DESCRIPTION:
Study Description:

We hypothesize that primary sclerosing cholangitis (PSC) develops as a consequence of a genetically driven aberrant immune response to commensal or pathogenic bacteria, and that unique genetic-immunemicrobial associations may underlie development of distinct disease patterns. We intend to conduct a thorough radiologic, endoscopic, histologic and microbiological investigation of patients with PSC in order to determine potential associations.

Objectives:

Primary Objective:

The ultimate goal of this study is to generate understanding of how factors driving pathogenesis in PSC interact by capturing and integrating collated datasets from across relevant biologic systems and interpreting those in the context of phenotypic presentation in one exceptionally well-characterized set of patients.

Secondary Objectives:

1. To collect comprehensive data on distinct patterns of disease expression, through single cell sequencing and microRNA and transcriptome profiling.
2. To conduct extensive phenotypic characterization of cellular and humoral immune responses as well as microbiome signatures at multiple anatomic sites.
3. To evaluate metabolic signatures or biomarkers for PSC diagnosis and prognostication.
4. To generate a humanized mouse model of each subject s disease by obtaining bone marrow aspirate.

Endpoints:

Primary Endpoint:

1. Identification of immune signatures at multiple levels and from different anatomical sites and tissues
2. Characterization of microbiome signatures (taxonomic and functional), as well as identification of specific species.
3. Identification of metabolomic signatures from different anatomical sites and tissues as well as identification of different biomarkers correlating with disease progression.
4. MicroRNA profiling of portal and systemic blood.

ELIGIBILITY:
* PSC SUBJECTS:

INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or nonpregnant female, greater than or equal to 18 years of age
3. Evidence of PSC established by biochemical testing and either MRCP or ERCP. Participant must have evidence of large duct disease on imaging.
4. Agreement to adhere to Lifestyle Considerations throughout study duration.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnant or lactating women or females of child-bearing age not taking measures to prevent pregnancy during the period of study.
2. History of clinical, serologic, or histopathologic evidence supporting etiologies of chronic liver disease other than PSC
3. History of liver transplantation
4. Diagnosis consistent with secondary sclerosing cholangitis (cholelithiasis, bile duct strictures secondary to ischemia, HIV cholangiopathy, etc.).
5. Current or past clinical evidence of decompensated liver disease (e.g. ascites, bleeding esophageal varices, spontaneous bacterial peritonitis, encephalopathy, etc.).
6. History of liver or bile duct lesions concerning for malignancy.
7. Ca-19-9 >130 U/microL
8. Alpha-fetoprotein level greater than 200 ng/microL.
9. Patients with active bacterial, viral, or fungal, systemic or localized infection.
10. Unwillingness to refrain from ingesting probiotics during study.
11. History of systemic disease not related to PSC that is poorly controlled or associated with declining functional status. Examples include but are not limited to: poorly controlled diabetes mellitus, chronic renal failure with eGFR is <60 microl/min/1.73m^2, chronic

    symptomatic heart failure or severe COPD.
12. Patients with history of any gastrointestinal malignancy in the last 3 years prior to enrollment will be excluded. Patients with history of any malignancy in the last 3 years prior to enrollment other than those individuals who had undergone curative surgical therapy and deemed as low risk for recurrence by her/his treating physician would be excluded.
13. History of portal vein thrombosis
14. Patients with severe allergic reactions to iodine or other contrast, which cannot be controlled by premedication with antihistamines or steroids.
15. History of gastric and/or proximal small bowel surgery including bariatric surgery such as Roux-en-Y gastric bypass
16. Contraindication to monitored anesthesia care and/or medications that are commonly used for conscious sedation during GI Endoscopy
17. Use of anti-coagulant and anti-platelet agents excluding aspirin and NSAIDs
18. Contraindications to completing MRCP or MRI
19. Absolute neutrophil count below 1000/mm^3
20. Hemoglobin level below 10.0 g/dl
21. Platelet count lower than 50,000/mm^3.
22. INR greater than or equal to 1.5, PTT greater thna or equal to 1.3 times control and/or any known history of disease associated with

    increased bleeding diathesis.
23. Inability to provide informed consent

CONTROLS:

INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female greater than or equal to 18 years of age
2. Any individual who is either a parent, sibling or child of a PSC patient enrolled to the study, or an unrelated person who has been living with the patient for at least 3 consecutive months before study enrollment

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History suggestive of PSC
2. History of chronic liver disease (except for steatosis)
3. Patients with history of any malignancy in the last 3 years prior to enrollment other than those individuals who had undergone curative surgical therapy and deemed as low risk for recurrence by her/his treating physician would be excluded.
4. History of Inflammatory Bowel Disease
5. Antibiotic use within the last 6 weeks
6. Pregnancy
7. Inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 male and female adult patients 18 years of age or above with known PSC recruited from hospitals in the continental US. 90 healthy volunteers, male and female 18 years of age or above, who are either family members of participating patients with PSC or have been cohabitating with participating patients with PSC.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The ultimate goal of this study is to generate understanding of how factors driving pathogenesis in PSC interact by capturing and integrating collated datasets from across relevant biologic systems and interpreting those in the context of phenot... | End of Study
  1. Identification of immune signatures at multiple levels and from different anatomical sites and tissues 2. Characterization of microbiome signatures (taxonomic and functional), as well as identification of specific species. 3. Identification of metabolomic signatures from different anatomical sites and tissues as well as identification of different biomarkers correlating with disease progression. 4. MicroRNA profiling of portal and systemic blood.

SECONDARY OUTCOMES:
To collect comprehensive data on distinct patterns of disease expression, through single cell sequencing and microRNA and transcriptome profiling. | End of Study
  Single cell sequencing, microRNA and transcriptome profiling
To conduct extensive phenotypic characterization of cellular and humoral immune responses as well as microbiome signatures at multiple anatomic sites | End of Study
  Immune phenotyping, immune repertoire sequencing and cytokine profiling techniques, as well as next generation sequencing of microbiota in saliva, stool, blood, bile, small intestine, colon and liver tissue
To evaluate metabolic signatures or biomarkers for PSC diagnosis and prognostication | End of Study
  High throughput metabolomics screening of portal and systemic blood, liver tissue and bile in search of bile acids and other target metabolites
To generate a humanized mouse model of each subject s disease by obtaining bone marrow aspirate | End of Study
  The study of immune phenotype and function in a host (in this case the mouse) na(SqrRoot) ve to immunosuppressive therapy

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000130-DK.html